CLINICAL TRIAL: NCT00194129
Title: A Randomized, Double Blind Comparison of Lithium Monotherapy Versus Lithium Plus Divalproex for the Outpatient Management of Hypomania/Mania in Patients With Rapid Cycling Bipolar Disorder Comorbid With Substance Abuse/Dependence
Brief Title: Lithium and Divalproex for the Treatment of Comorbid Rapid Cycling Bipolar Disorder and Substance Abuse Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Abbott (Industry)
Responsible Party: Principal Investigator, Joseph Calabrese, MD, Director, Mood Disorders Program, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH050165 (NIH); R01MH050165 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Lithium Carbonate; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium plus Divalproex (Experimental): Patients assigned to the combination group were continued on lithium and blinded divalproex.
  Interventions: Drug: Lithium; Drug: Divalproex
- Lithium plus placebo (Placebo Comparator): Patients assigned to lithium monotherapy underwent divalproex-placebo substitution at a rate of 250 mg decrements every week until discontinued.
  Interventions: Drug: Lithium; Drug: Placebo

INTERVENTIONS:
Drug: Lithium — Lithium monotherapy was initiated at 300 mg twice daily and titrated over 3-6 weeks to minimum blood levels of 0.8 meq/L.
  Other Names: Lithium Carbonate
Drug: Divalproex — Divalproex was then initiated at 250 mg twice daily and increased over 3-6 weeks to minimum blood levels of 50 ug/ml.
  Other Names: Valproic Acid; Depakote
  Arms: Lithium plus Divalproex
Drug: Placebo — Placebo pills that looked exact to divaloproex were provided to subjects and take twice daily.
  Arms: Lithium plus placebo

SUMMARY:
This study will determine the efficacy and safety of combination therapy with divalproex and lithium for treating mania in people with rapid cycling bipolar disorder and a substance abuse disorder.

DETAILED DESCRIPTION:
Longitudinal Evaluation of the Efficacy and Safety of Divalproex and Lithium in Dual Diagnosis Bipolar Rapid Cycling: This study recruits males and females age 18 and older who currently meet diagnostic criteria for rapid cycling bipolar disorder (type I or II) and who have met the criteria for substance abuse or dependence of cocaine, marijuana and/or alcohol within the past six months. Patients are initially stabilized on dual therapy of lithium and depakote and then randomly assigned to double-blind treatment with either lithium monotherapy or continued dual therapy. Patients remain in the study for six months or until they experience a relapse. Patients in this study are required to bring a friend or family member to all study visits as well as attend chemical dependency services. This study is sponsored by the NIMH. Subjects receive study-related care at no cost.

ELIGIBILITY:
Inclusion Criteria:

* To be included in this study, patients will be required to be either acutely hypomanic or manic as defined by the Diagnostic and Statistical Manual -IV (DSM-IV) and meet criteria for current substance abuse and/or dependence disorder within the last six months.
* Must have 4 or more episodes in the immediate 12 months prior to study entry.
* Males or females 16 - 65 years of age.
* A score of 60 or less on the Global Assessment Scale.
* Have no medical illness precluding the use of lithium or divalproex.

Exclusion Criteria:

* Patients who have had intolerable side effects to lithium levels 0.8 meq/L or divalproex levels of 50 ug/ml. Patients who have been completely non-responsive to lithium in the past will be excluded, whereas patients who have had partial responses to lithium will be permitted into the study.
* Patients with a prior history of seizure disorder, cerebral vascular disease, structural brain damage from trauma, clinically significant focal neurological abnormalities, EEG abnormalities with frank paroxysmal activity or a previous CT/MRI scan of the brain with gross structural abnormalities.
* Patients who require anticoagulant drug therapy.
* Patients who have uncontrolled gastrointestinal, renal, hepatic, endocrine, cardiovascular, pulmonary, immunological or hematological disease. Patients with alcohol-related liver disease as reflected by diffuse elevations in liver functions tests exceeding the upper limits of the normal range by 50% will be excluded.
* Patients who are pregnant or plan to become pregnant during the study.
* Patients who have received haloperidol decanoate or fluphenazine decanoate within the last 10 weeks.
* Patients who have a central nervous system (CNS) neoplasm, uncontrolled metabolic, demyelinating or progressive disorder; active CNS infection; or any progressive neurological disorder.
* Patients who are taking exogenous steroids.
* Patients who do not meet criteria for substance abuse or dependence.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 1997-11; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Calabrese, MD, Principal Investigator — Case Western Reserve University / University Hospitals of Cleveland
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Kemp DE, Gao K, Ganocy SJ, Elhaj O, Bilali SR, Conroy C, Findling RL, Calabrese JR. A 6-month, double-blind, maintenance trial of lithium monotherapy versus the combination of lithium and divalproex for rapid-cycling bipolar disorder and Co-occurring substance abuse or dependence. J Clin Psychiatry. 2009 Jan;70(1):113-21. doi: 10.4088/jcp.07m04022. Epub 2008 Dec 30. PMID 19192457
- [Derived] Gao K, Verduin ML, Kemp DE, Tolliver BK, Ganocy SJ, Elhaj O, Bilali S, Brady KT, Findling RL, Calabrese JR. Clinical correlates of patients with rapid-cycling bipolar disorder and a recent history of substance use disorder: a subtype comparison from baseline data of 2 randomized, placebo-controlled trials. J Clin Psychiatry. 2008 Jul;69(7):1057-63. doi: 10.4088/jcp.v69n0703. PMID 18588360

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at the outpatient Mood Disorders Program of Case Western Reserve University/University Hospitals Case Medical Center between October 1997 and October 2006.
Pre-assignment Details: Patients meeting stabilization criteria for a minimum of 4 consecutive weeks were eligible for random assignment to double-blind maintenance treatment. Patients not meeting these criteria by 24 weeks were discontinued from the study.
Groups:
- Lithium Plus Divalproex: Participants were given lithium monotherapy was initiated at 300 mg twice daily and titrated over 3-6 weeks to minimum blood levels of 0.8 meq/L. If randomized to divalproex arm, divalproex was then initiated at 250 mg twice daily and increased over 3-6 weeks to minimum blood levels of 50 ug/ml.
- Lithium Plus Placebo: Participants were given lithium monotherapy was initiated at 300 mg twice daily and titrated over 3-6 weeks to minimum blood levels of 0.8 meq/L. If randomized to placebo arm, placebo pills that looked exact to divaloproex were provided to subjects and take twice daily.
Period: Overall Study
Arm/Group | Lithium Plus Divalproex | Lithium Plus Placebo
Started | 15 | 16
Completed | 5 | 3
Not Completed | 10 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium Plus Divalproex | Lithium Plus Placebo | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (10.9) | 40 (10.6) | 38.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 9 | 12 | 21
Illness Type [Number; unit: participants] — Bipolar I disorder involves periods of severe mood episodes from mania to depression. Bipolar II disorder is a milder form of mood elevation, involving milder episodes of hypomania that alternate with periods of severe depression.
  participants
    Bipolar I disorder | 13 | 13 | 26
    Bipolar II disorder | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment for Emerging Symptoms of a Mood Relapse
Description: A relapse is a return to either a depressive, manic, hypomanic or mixed episode after a period of not have any symptoms.
Time Frame: Up to 6 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lithium Plus Divalproex | Lithium Plus Placebo
Number analyzed (Participants) | 15 | 16
weeks | 17.8 [12.8 to 27.6] | 15.9 [11.0 to 22.9]

2. Secondary Outcome: Time to Treatment for Emerging Symptoms of a Manic/Hypomanic/Mixed Episode
Time Frame: Up to 6 months
Population: Due to the heavily censored nature of this data, the median survival for time to treatment for emerging manic/hypomanic/mixed symptoms in both arms is not evaluable. Statistics software was unable to analyze the data.
Arm/Group | Lithium Plus Divalproex | Lithium Plus Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Treatment for Emerging Symptoms of a Depressive Episode
Time Frame: Up to 6 months
Population: Due to the heavily censored nature of this data, the median survival for time to treatment for emerging depression symptoms in both arms is not evaluable. Statistics software was unable to analyze the data.
Arm/Group | Lithium Plus Divalproex | Lithium Plus Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Rate of Alcohol Use Disorders After Open-label Treatment With Lithium and Divalproex
Description: Number of subjects who no longer met criteria for active abuse or had entered into early full remission after receiving up to 6 months of open-label treatment with lithium and divalproex
Time Frame: Baseline to Month 6
Population: This only includes subjects who had an alcohol use disorder at study entry. The purpose of this analysis was to see if treatment with both open-label lithium and divalproex during the first phase of study participation (i.e. prior to randomization to lithium monotherapy or continued dual therapy) lead to a change in rates of alcohol use disorders.
Measure: Count of Participants; unit: Participants
Groups:
- Completers: This analysis only includes subjects who had an alcohol use disorder at study entry.
Arm/Group | Completers
Number analyzed (Participants) | 19
Participants | 11

5. Secondary Outcome: Change in Rate of Cannabis Use Disorders After Open-label Treatment With Lithium and Divalproex
Description: Number of subjects who no longer met criteria for active cannabis abuse or had entered into early full remission after receiving up to 6 months of open-label treatment with lithium and divalproex
Time Frame: Baseline to Month 6
Population: This only includes subjects who had a cannabis use disorder at study entry. The purpose of this analysis was to see if treatment with both open-label lithium and divalproex during the first phase of study participation (i.e. prior to randomization to lithium monotherapy or continued dual therapy) lead to a change in rates of cannabis use disorders.
Measure: Count of Participants; unit: Participants
Groups:
- Completers: This only includes subjects who had a cannabis use disorder at study entry.
Arm/Group | Completers
Number analyzed (Participants) | 15
Participants | 8

6. Secondary Outcome: Change in Rate of Cocaine Use Disorders After Open-label Treatment With Lithium and Divalproex
Description: Number of subjects who no longer met criteria for active cocaine abuse or had entered into early full remission after receiving up to 6 months of open-label treatment with lithium and divalproex
Time Frame: Baseline to Month 6
Population: This only includes subjects who were using cocaine at the time of study entry. The purpose of this analysis was to see if treatment with both open-label lithium & divalproex during the first phase of study participation (i.e. prior to randomization to lithium monotherapy or continued dual therapy) lead to a change in rates of cocaine use disorders.
Measure: Count of Participants; unit: Participants
Groups:
- Completers: This only includes subjects who had cocaine use disorder at study entry.
Arm/Group | Completers
Number analyzed (Participants) | 9
Participants | 7

ADVERSE EVENTS:
Arm/Group | Lithium Plus Divalproex | Lithium Plus Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 13/15 | 13/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Plus Divalproex (N=15) | Lithium Plus Placebo (N=16)
Tremors (Nervous system disorders) | 10 (10) | 10 (10)
Polyuria/Polydipsia (Renal and urinary disorders) | 6 (6) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 6 (6)
Weight Gain (General disorders) | 2 (2) | 5 (5)
Fatigue (General disorders) | 5 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Alopecia (General disorders) | 3 (3) | 1 (1)
Dry Mouth (General disorders) | 3 (3) | 0 (0)
Sexual Dysfunction (Social circumstances) | 2 (2) | 2 (2)
Cognitive Dysfunction (Social circumstances) | 2 (2) | 2 (2)
Blurred Vision (Eye disorders) | 2 (2) | 1 (1)
Increased Appetite (General disorders) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No